CLINICAL TRIAL: NCT02829814
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study To Evaluate The EFFIcacy and Safety of TNX-102 SL Tablets Taken Daily At Bedtime In Patients With FibRoMyalgia
Brief Title: Repeat of: A Study to Evaluate Efficacy and Safety of Sublingual TNX-102 SL Tablet Taken at Bedtime in Patients With Fibromyalgia
Acronym: RE-AFFIRM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For business reason unrelated to safety or tolerability,Tonix discontinued this study.
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F302
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia; Myofascial Pain Syndromes; Muscular Diseases; Nervous System Diseases; Neuromuscular Diseases; Rheumatic Diseases; Musculoskeletal Diseases
Keywords: Pain; Sleep; Fibromyalgia; FM
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes; Muscular Diseases; Nervous System Diseases; Neuromuscular Diseases; Rheumatic Diseases; Musculoskeletal Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNX-102 SL Tablet, 2.8 mg (Experimental): 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 12 weeks
  Interventions: Drug: TNX-102 SL Tablet, 2.8 mg
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL Tablet, 2.8 mg — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablet, 2.8 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
The present trial is designed to assess the safety and efficacy of TNX-102 SL 2.8 mg tablets, taken daily at bedtime after 12 weeks of treatment in patients with fibromyalgia.

The use of low-dose sublingual formulation of cyclobenzaprine (TNX-102 SL) dosed nightly for fibromyalgia is supported by the results of TNX-CY-F202 Phase 2b study -- the results provide strong evidence that TNX-102 SL 2.8 mg dosed nightly results in beneficial effects upon pain, sleep and other FM symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Fibromyalgia (2010 ACR criteria)
* Male or female 18-75 years old
* Patients currently receiving pharmacologic treatment for depression should have been clinically stable for at least 3 months prior to randomization, and on stable doses of antidepressants during this 3 month time frame.
* Willing and able to withdraw specific therapies (ask PI)
* If female, medically acceptable form of contraception or not of child bearing potential.
* Provide written informed consent to participate.
* Willing and able to comply with all protocol specified requirement.

Exclusion Criteria:

* Arthritis, lupus and other systemic auto-immune diseases
* Regional or persistent pain that could interfere with assessment of fibromyalgia pain
* Bipolar and psychotic disorders
* Increased risk of suicide
* Significant clinical (cardiac, systemic infection, systemic corticosteroid requirement, drug/alcohol abuse) or laboratory abnormalities.
* Inability to wash-out specific medications (ask PI)
* Known hypersensitivity to cyclobenzaprine
* Others: seizure disorders, severe/untreated sleep apnea, BMI>45

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Oceanside, California
  - San Diego, California
  - Brandon, Florida
  - DeLand, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Jackson, Mississippi
  - Las Vegas, Nevada
  - Cedarhurst, New York
  - Williamsville, New York
  - Raleigh, North Carolina
  - Fargo, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Started | 27 | 24
Completed | 0 | 0
Not Completed | 27 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.10) | 52.1 (7.45) | 51.7 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are 2 patients in the placebo group for whom sex was not recorded.
  Participants
    number analyzed (Participants) | 25 | 24 | 49
    Female | 24 | 23 | 47
    Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Weekly Mean Pain Score
Description: The primary efficacy endpoint is the proportion of patients with a ≥30% improvement from baseline to Week 12 in the weekly average of the daily self-reported average pain severity score using an 11-point (0-10) numeric response scale (NRS). A score of 0 indicates "no pain at all", and a score of 10 indicates "worst possible pain".
Time Frame: Day 1, Week 12
Population: This study was stopped for business reasons prior to any patients completing the study. Therefore, no efficacy analyses were performed.
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: Proportion of patients with a PGIC rating of "very much improved" or "much improved" at Week 12.The PGIC is a 7-point scale (1=very much improved; 7=very much worse) that assesses the patient's perception of the overall change in his/her fibromyalgia symptoms since entering the study.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQR) Revised, Symptoms Domain
Description: Change from Baseline in the FIQR symptoms domain score at Week 12. The FIQ-R symptom domain is composed of 10 questions. All questions are based on an 11-point numerical rating scale (NRS) of 0-10, with 10 being "worst." Symptom domain scores range from 0-100, with higher scores reflecting worse status.
Time Frame: Day 1, Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQR) Revised, Functional Domain Score
Description: Change from Baseline in the FIQR function domain score at Week 12. The FIQ-R functional domain score is composed of 9 questions which are rated on an 11-point numerical rating scale (NRS) of 0-10, with 10 being "worst." FIQ-R functional domain scores can range from 0-90, with higher scores reflecting worsening status.
Time Frame: Day 1, Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Daily Diary Sleep
Description: Change from Baseline in the weekly average of the daily diary assessment of sleep quality at Week 12. Daily sleep quality was measured using an 11-point (0-10) numerical rating scale (NRS), with higher scores representing worse sleep.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Reported Outcomes Measurement System (PROMIS), Sleep Disturbance
Description: Change from Baseline in the PROMIS score for sleep disturbance at Week 12. The Patient-Reported Outcome Measurement Information System (PROMIS) sleep disturbance instrument consists of 8 items in which responses are scored 1 to 5 for each item. PROMIS scores are presented as T-scores in which the raw score has been rescaled into a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores represent more of the concept being measured (in this case, sleep disturbance).
Time Frame: Day 1, Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient Reported Outcomes Measurement System (PROMIS), Fatigue
Description: Change from Baseline in the PROMIS score for fatigue at Week 12. The Patient-Reported Outcome Measurement Information System (PROMIS) fatigue instrument consists of 8 items in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores are first synchronized prior to calculation of the total raw score. PROMIS scores are presented as T-scores in which the raw score has been rescaled into a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores represent more of the concept being measured (in this case, sleep disturbance).
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Daily Diary Pain
Description: Change from baseline to Week 12 in the weekly average of the daily self-reported average pain severity score. Average daily pain was measured using an 11-point (0-10) numerical rating scale (NRS), with higher scores representing worse pain. Weekly averages were calculated based on the reported daily scores.
Time Frame: Week -1 (Day -7 to Day -1), Week 12
Population: as for outcome 1
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 7 weeks
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.